CLINICAL TRIAL: NCT02276859
Title: The Optimal Type of Bolus Following a High-protein Meal in Type 1 Diabetic Children Treated With Insulin Pumps
Brief Title: Normal Versus Dual Wave Insulin Bolus for High-protein Food
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Protein Food Insulin Bolus
Record Dates: First submitted 2014-10-07; First posted 2014-10-28 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2014-09

CONDITIONS: Type 1 Diabetes
Keywords: dual-wave bolus; square bolus; normal bolus; standard bolus; high-protein meal; prandial insulin requirement
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; Insulin Lispro; insulin glulisine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal/ Dual-wave (Experimental): On the first study day, pre-breakfast insulin was given as a normal bolus 15 minutes before a standardized high-protein meal. On the second day, pre-breakfast insulin was given as a dual-wave bolus before the same high-protein meal.
  The carbo-insulin and fat-protein-insulin ratio on both study days were identical to the patient's ratio when entering trial.
  Kind of study bolus insulin will be a rapid-acting insulin analog same as previously used by the participant (before entering the trial) - insulin aspart, insulin lispro or insulin glulisine
  Interventions: Drug: insulin aspart; Drug: insulin lispro; Drug: insulin glulisine
- Dual-wave/Normal (Experimental): On the first study day, pre-breakfast insulin was given as a dual-wave bolus 15 minutes before a standardized high-protein meal. On the second day, pre-breakfast insulin was given as a normal bolus before the same high-protein meal.
  The carbo-insulin and fat-protein-insulin ratio on both study days were identical to the patient's ratio when entering trial.
  Kind of study bolus insulin will be a rapid-acting insulin analog same as previously used by the participant (before entering the trial) - insulin aspart, insulin lispro or insulin glulisine
  Interventions: Drug: insulin aspart; Drug: insulin lispro; Drug: insulin glulisine

INTERVENTIONS:
Drug: insulin aspart — A kind of study bolus insulin will be insulin aspart if participant used insulin aspart before entering the trial
  Other Names: NovoRapid®
Drug: insulin lispro — A kind of study bolus insulin will be insulin lispro if participant used insulin lispro before entering the trial
  Other Names: Humalog®
Drug: insulin glulisine — A kind of study bolus insulin will be insulin glulisine if participant used insulin glulisine before entering the trial
  Other Names: Apidra®

SUMMARY:
Patients receive a standardized high-protein test meal at breakfast time. Insulin is given as bolus (normal or dual-wave (normal plus square) and basal rate using an insulin pump. The 3h post-meal glucose excursions will be recorded by self-blood glucose measurements (SMBG) (every 1 hour) and continuous glucose monitoring system (CGMS). The intervention is taking part under in-patient clinical conditions.

DETAILED DESCRIPTION:
The dual-wave bolus delivers an immediate normal pre-meal insulin bolus followed by square-wave bolus that is evenly delivered over several hours as programmed by the patient. The aim of this study is to compare post-prandial glycaemic excursions following a high-protein meal after administration of insulin by normal vs dual-wave bolus. During this prospective, cross-over, repeated measures study, pediatric patients with type 1 diabetes, treated with insulin pump therapy will be evaluated using the self-blood glucose measurements following standardized high-protein meal and two types of boluses (normal or dual-wave). The required insulin dose will be calculated based on patient's insulin-exchange ratio. A high-protein meal will be given on two subsequent breakfasts and comparisons will be made between normal and dual-wave insulin bolus delivery. Prolonged post-prandial glycaemic excursions will be identified using the CGMS.

ELIGIBILITY:
Inclusion Criteria:

* duration of type 1 diabetes longer than 12 months
* insulin pump therapy longer than 3 months
* written informed consent by patients and parents
* patients must be willing to wear a glucose sensor for two days
* insulin requirement more than 0,5 units/kg/day

Exclusion Criteria:

* concomitant dietary restrictions (e.g. celiac disease or food allergy)
* diabetes related complications (e.g. nephropathy)
* any disease judged by the investigator to affect the trial
* withdrawal of consent to participate in the study

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemia | 60 minutes after the meal
  Post-prandial blood glucose excursions measured by self monitoring of blood glucose (SMBG)
Postprandial glycemia | 120 minutes after the meal
  Post-prandial blood glucose excursions measured by self monitoring of blood glucose
Postprandial glycemia | 180 minutes after the meal
  Post-prandial blood glucose excursions measured by self monitoring of blood glucose

SECONDARY OUTCOMES:
Hypoglycemia episodes | 3-hour study period
  Hypoglycemia defined as a plasma glucose concentration below 65 mg/dl with or without symptoms
Glucose Area Under the Curve (AUC) | 3-hour study period
  measurements based on CGMS
Mean amplitude of glycemic excursion | 3-hour study period
  measurements based on CGMS

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Szypowska, Study Chair — University of Alberta; Katarzyna Piechowiak, Principal Investigator — University of Alberta
Locations (1):
- Department of Pediatrics, Medical University of Warsaw, Poland, Warsaw, Poland